CLINICAL TRIAL: NCT03263663
Title: Optimization of Individualized Therapy for CRCs With Secondary RESISTance Towards Anti-EGFR Targeted Therapy Using an Avatar Model (Colon-Resist-Net)
Brief Title: Optimization of Individualized Therapy for CRCs With Secondary RESISTance Towards Anti-EGFR Targeted Therapy Using an Avatar Model
Acronym: 2016-003295-46
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: MGO Ruhr-University Bochum (RUB) (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Director of the CCC LMU, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: RESIST
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Colo-rectal Cancer; RAS Wild-type; UICC III; UICC II + RF; UICC IV Curative Intent
Keywords: colorectal cancer; adjuvant
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary tumormaterial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chemotherapy plus targeted treatment: Patients are treated in second-line with chemotherapy plus a targeted treatment according to the resistance mechanism to cetuximab pretreatment
  Interventions: Drug: targeted substance according to the avatar model
- Chemotherapy according to physician choice standard: Patients are treated in second-line with chemotherapy according to physicians choice after cetuximab pretreatment

INTERVENTIONS:
Drug: targeted substance according to the avatar model — individualized second line treatment
  Groups: Chemotherapy plus targeted treatment

SUMMARY:
In this exploratory phase II trial, the possibility of a personalized treatment after resistance to cetuximab will be evaluated. Therefore, tumor material of all patients shall be obtained, transferred into avatars and treated the same way as in the patient until resistance arises. These resistant tumor cells are subsequently treated by different targeted treatment combinations in the mouse avatar model to find the most active drug or combination of drugs. This drug or combination of drugs may then be offered to the patient after cetuximab resistance has occurred. Multiple liquid biopsies shall be obtained in patients during first-line treatment with cetuximab as well as during second line experimental treatment to monitor mutations that may be associated with cetuximab resistance. Furthermore at the time of resistance a biopsy should be taken and analyzed to ensure that the mechanism of resistance seen in the avatar model matches with the mechanism of resistance in the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age ≥ 18 years
* Written declaration of consent
* ECOG Performance Status 0-1
* Life expectancy> 3 months
* Histologically confirmed adenocarcinoma of the colon or rectum at stage UICC III or UICC IV
* Histologically confirmed adenocarcinoma of the colon or rectum in stage UICC II with one of the following risk factors: CEA> 200; T4 tumor, emergency surgery, <12 distant lymph nodes, surgery due to intestinal obstruction (ileus)
* Patient agrees to the preservation of tumor material for the purpose of molecular analyzes including the determination of the genetic profile of the tumor (participation in the project "RESIST")

Exclusion Criteria:

* Preoperative Radiotherapy
* Preoperative chemotherapy
* Heart failure> Grade II (functional NYHA classification)
* Existing concomitant disease or condition that would make the patient unsuitable for a study participation or interfere with the safety of the subject
* Any psychological, familial, sociological or geographical event which does not allow observance of the study protocol
* Additional carcinoma therapy (chemotherapy, radiation, biological therapy, immunotherapy or hormonal therapy) during the study
* Known malignant second neoplasia within the last 5 years (except for a basal cell carcinoma or a carcinoma in situ of the uterine cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced colorectal cancer
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free-survival | 5-7 months
  according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Stintzing, Prof. Dr., Principal Investigator — Senior Physician
Locations (1):
- University of Munich - Klinikum der Universitaet Muenchen, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes